CLINICAL TRIAL: NCT00395161
Title: The Critical Illness Stress-induced Immune Suppression Prevention Trial
Brief Title: The CRISIS Prevention Study
Acronym: CRISIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated for futility on 11/30/09 based on the recommendation of the DSMB
Sponsor: Michael Dean (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Seattle Children's Hospital (Other); Children's Hospital Los Angeles (Other); Arkansas Children's Hospital Research Institute (Other); Children's Hospital of Michigan (Other); University of Pittsburgh (Other); Children's National Research Institute (Other); University of California, Los Angeles (Other); Harborview Injury Prevention and Research Center (Other)
Responsible Party: Sponsor-Investigator, Michael Dean, Data Coordinating Center Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01HD049934 (NIH)
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Sepsis
Keywords: sepsis; prevention; mineral supplementation
MeSH Terms: conditions — Sepsis | interventions — Metoclopramide; Zinc; Glutamine; Selenium; Sodium Chloride; Whey

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zinc selenium glutamine metoclopramide (Experimental): metoclopramide, zinc, selenium, and glutamine
  Interventions: Drug: Metoclopramide; Drug: Zinc; Dietary Supplement: Glutamine; Drug: Selenium
- enteral whey protein and IV saline (Placebo Comparator): saline, sterile water, whey protein
  Interventions: Other: saline; Other: sterile water; Other: selenium; Dietary Supplement: whey-protein

INTERVENTIONS:
Drug: Metoclopramide — 0.2 mg/kg/dose IV every 12 hours
  Other Names: Reglan
  Arms: zinc selenium glutamine metoclopramide
Drug: Zinc — one enteral dose daily of zinc chloride (10 mg/day elemental zinc for infants < or equal to one year of age, and 20 mg/day elemental zinc for patients > 1 year of age)
  Arms: zinc selenium glutamine metoclopramide
Dietary Supplement: Glutamine — one enteral dose daily of glutamine 0.3 gm/kg/day
  Arms: zinc selenium glutamine metoclopramide
Drug: Selenium — one enteral dose daily of selenium (40 μg for infants < 8 months of age, 60 μg for infants 8 to 12 months of age, 90 μg for children 1-3 years, 150 μg for children 4-8 years, 280 μg for children 9 to 13 years, and 400 μg for children > 13 years)
  Arms: zinc selenium glutamine metoclopramide
Other: saline — equivalent volume of intravenous saline
  Arms: enteral whey protein and IV saline
Other: sterile water — equivalent volume of sterile water
  Arms: enteral whey protein and IV saline
Other: selenium — equivalent volume of sterile water
  Arms: enteral whey protein and IV saline
Dietary Supplement: whey-protein — one enteral dose daily of whey-protein
  Other Names: Beneprotein
  Arms: enteral whey protein and IV saline

SUMMARY:
Despite strict hand washing, sterile technique, and antibiotic-coated catheters, nosocomial infection and sepsis remain the leading acquired causes of morbidity and mortality in critically ill children. Subsequent use of antibiotics to treat nosocomial infection and sepsis is considered a major attributable factor in the rise of antibiotic-resistant organisms in this population of children. This study will use a double-blind, randomized, controlled trial design to test the hypothesis that daily prophylaxis with metoclopramide, zinc, selenium and glutamine will reduce nosocomial infection and sepsis in critically ill children.

DETAILED DESCRIPTION:
Despite strict hand washing, sterile technique, and antibiotic-coated catheters, nosocomial infection and sepsis remain the leading acquired causes of morbidity and mortality in critically ill children. Subsequent use of antibiotics to treat nosocomial infection and sepsis is considered a major attributable factor in the rise of antibiotic-resistant organisms in this population of children. Presently, "prophylaxis" strategies are used to prevent stress-induced gastrointestinal bleeding; however, no "prophylaxis" strategy is used to prevent stress-induced nosocomial infection and sepsis. When left unopposed, the stress hormone, cortisol, induces lymphocyte apoptosis, lymphopenia, and immune insufficiency. Prolactin is the counter-regulatory stress hormone that prevents cortisol-induced apoptosis and immunosuppression. Zinc, selenium, and glutamine are also important in maintenance of lymphocyte health. Critically ill patients commonly develop hypoprolactinemia secondary to increased central nervous system dopaminergic activity, as well as zinc, selenium, and glutamine deficiency caused by increased utilization and decreased supply. Hypoprolactinemia can be prevented by metoclopramide, a dopamine 2 receptor antagonist commonly used as a prokinetic in children, and zinc, selenium, and glutamine deficiency can be prevented with enteral supplementation. This study will use a double-blind randomized controlled trial design to test the hypothesis that daily prophylaxis with metoclopramide, zinc, selenium and glutamine will reduce nosocomial infection and sepsis in critically ill children.

ELIGIBILITY:
Inclusion Criteria:

During the initial accrual period for this study, prior to the first interim analysis, patients will be eligible for enrollment if they:

* are between 12 months and less than 18 years; AND
* are within the first 48 hours of the PICU admission; AND
* have an endotracheal tube, central venous catheter (new or old, tunneled or not tunneled), or Foley catheter; AND
* are anticipated to have an indwelling arterial or central venous catheter for blood sampling during the first three days of study enrollment.

After the Data Safety Monitoring Board (DSMB) conducts its first interim evaluation, after enrollment of approximately 200 subjects, a decision will be made by the DSMB concerning enrollment of subjects between 40 weeks gestational age and 12 months. If the DSMB approves enrollment of infants after the first interim analysis, then patients will be eligible for enrollment if they:

* are between 40 weeks gestational age and less than 18 years; AND
* are within the first 48 hours of the PICU admission; AND
* have an endotracheal tube, central venous catheter (new or old, tunneled or not tunneled), or Foley catheter; AND
* are anticipated to have an indwelling arterial or central venous catheter for blood sampling during the first three days of study enrollment.

Exclusion Criteria:

During the initial accrual period for this study, prior to the first interim analysis, patients will be ineligible for enrollment if ANY of the following is true or anticipated:

* are less than 1 year age; OR
* are greater than or equal to 18 years of age; OR
* have a known allergy to metoclopramide; OR
* planned removal of endotracheal tube, central venous catheter, AND Foley catheters, within 72 hours of study enrollment, OR
* suspected intestinal obstruction, OR
* intestinal surgery or bowel disruption, OR
* chronic metoclopramide therapy prior to enrollment, OR
* failure to enroll within 48 hours of PICU admission, OR
* readmission to PICU in the previous 28 days, OR
* previously enrolled in this study, OR
* lack of commitment to aggressive intensive care therapies.

After the Data Safety Monitoring Board (DSMB) conducts its first interim evaluation, after enrollment of approximately 200 subjects, a decision will be made by the DSMB concerning enrollment of subjects between 40 weeks gestational age and 12 months. If the DSMB approves enrollment of infants after the first interim analysis, then patients will be ineligible for enrollment if ANY of the following is true or anticipated:

* are less than 40 weeks gestational age; OR
* are greater than or equal to 18 years of age; OR
* have a known allergy to metoclopramide; OR
* planned removal of endotracheal tube, central venous catheter, AND Foley catheters, within 72 hours of study enrollment, OR
* suspected intestinal obstruction

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Carcillo, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Watson RS, Carcillo JA, Linde-Zwirble WT, Clermont G, Lidicker J, Angus DC. The epidemiology of severe sepsis in children in the United States. Am J Respir Crit Care Med. 2003 Mar 1;167(5):695-701. doi: 10.1164/rccm.200207-682OC. Epub 2002 Nov 14. PMID 12433670
- [Background] Brown RB, Stechenberg B, Sands M, Hosmer D, Ryczak M. Infections in a pediatric intensive care unit. Am J Dis Child. 1987 Mar;141(3):267-70. doi: 10.1001/archpedi.1987.04460030045021. PMID 3812407
- [Background] Stein F, Trevino R. Nosocomial infections in the pediatric intensive care unit. Pediatr Clin North Am. 1994 Dec;41(6):1245-57. doi: 10.1016/s0031-3955(16)38871-x. PMID 7984384
- [Background] Ford-Jones EL, Mindorff CM, Pollock E, Milner R, Bohn D, Edmonds J, Barker G, Gold R. Evaluation of a new method of detection of nosocomial infection in the pediatric intensive care unit: the Infection Control Sentinel Sheet System. Infect Control Hosp Epidemiol. 1989 Nov;10(11):515-20. doi: 10.1086/645938. PMID 2685101
- [Background] Milliken J, Tait GA, Ford-Jones EL, Mindorff CM, Gold R, Mullins G. Nosocomial infections in a pediatric intensive care unit. Crit Care Med. 1988 Mar;16(3):233-7. doi: 10.1097/00003246-198803000-00005. PMID 3277780
- [Background] Allen U, Ford-Jones EL. Nosocomial infections in the pediatric patient: an update. Am J Infect Control. 1990 Jun;18(3):176-93. doi: 10.1016/0196-6553(90)90183-s. PMID 2194407
- [Background] Donowitz LG. High risk of nosocomial infection in the pediatric critical care patient. Crit Care Med. 1986 Jan;14(1):26-8. doi: 10.1097/00003246-198601000-00006. PMID 3510104
- [Background] Meakins JL, Pietsch JB, Bubenick O, Kelly R, Rode H, Gordon J, MacLean LD. Delayed hypersensitivity: indicator of acquired failure of host defenses in sepsis and trauma. Ann Surg. 1977 Sep;186(3):241-50. doi: 10.1097/00000658-197709000-00002. PMID 142452
- [Background] Pellegrini JD, De AK, Kodys K, Puyana JC, Furse RK, Miller-Graziano C. Relationships between T lymphocyte apoptosis and anergy following trauma. J Surg Res. 2000 Feb;88(2):200-6. doi: 10.1006/jsre.1999.5797. PMID 10644489
- [Background] O'Sullivan ST, Lederer JA, Horgan AF, Chin DH, Mannick JA, Rodrick ML. Major injury leads to predominance of the T helper-2 lymphocyte phenotype and diminished interleukin-12 production associated with decreased resistance to infection. Ann Surg. 1995 Oct;222(4):482-90; discussion 490-2. doi: 10.1097/00000658-199522240-00006. PMID 7574928
- [Background] Menges T, Engel J, Welters I, Wagner RM, Little S, Ruwoldt R, Wollbrueck M, Hempelmann G. Changes in blood lymphocyte populations after multiple trauma: association with posttraumatic complications. Crit Care Med. 1999 Apr;27(4):733-40. doi: 10.1097/00003246-199904000-00026. PMID 10321662
- [Background] Gogos CA, Drosou E, Bassaris HP, Skoutelis A. Pro- versus anti-inflammatory cytokine profile in patients with severe sepsis: a marker for prognosis and future therapeutic options. J Infect Dis. 2000 Jan;181(1):176-80. doi: 10.1086/315214. PMID 10608764
- [Background] Rathmell JC, Thompson CB. Pathways of apoptosis in lymphocyte development, homeostasis, and disease. Cell. 2002 Apr;109 Suppl:S97-107. doi: 10.1016/s0092-8674(02)00704-3. PMID 11983156
- [Background] Fletcher-Chiappini SE, Compton MM, LaVoie HA, Day EB, Witorsch RJ. Glucocorticoid-prolactin interactions in Nb2 lymphoma cells: antiproliferative versus anticytolytic effects. Proc Soc Exp Biol Med. 1993 Mar;202(3):345-52. doi: 10.3181/00379727-202-43545. PMID 8437991
- [Background] Ayala A, Herdon CD, Lehman DL, DeMaso CM, Ayala CA, Chaudry IH. The induction of accelerated thymic programmed cell death during polymicrobial sepsis: control by corticosteroids but not tumor necrosis factor. Shock. 1995 Apr;3(4):259-67. doi: 10.1097/00024382-199504000-00003. PMID 7600193
- [Background] Tarcic N, Ovadia H, Weiss DW, Weidenfeld J. Restraint stress-induced thymic involution and cell apoptosis are dependent on endogenous glucocorticoids. J Neuroimmunol. 1998 Feb;82(1):40-46. doi: 10.1016/S0165-5728(97)00186-0. PMID 9526844
- [Background] Noel GL, Suh HK, Stone JG, Frantz AG. Human prolactin and growth hormone release during surgery and other conditions of stress. J Clin Endocrinol Metab. 1972 Dec;35(6):840-51. doi: 10.1210/jcem-35-6-840. No abstract available. PMID 4634485
- [Background] Yu-Lee LY. Molecular actions of prolactin in the immune system. Proc Soc Exp Biol Med. 1997 May;215(1):35-52. doi: 10.3181/00379727-215-44111. PMID 9142136
- [Background] Freeman ME, Kanyicska B, Lerant A, Nagy G. Prolactin: structure, function, and regulation of secretion. Physiol Rev. 2000 Oct;80(4):1523-631. doi: 10.1152/physrev.2000.80.4.1523. PMID 11015620
- [Background] L Vankrieken. Immulite reproductive hormone assays: multicenter reference range data, 2000.
- [Background] HG Friesen. Human prolactin. Ann Rev Coll Phys Surg Can, 11:275- 281, 1978.
- [Background] Buckley AR, Buckley DJ. Prolactin regulation of apoptosis-associated gene expression in T cells. Ann N Y Acad Sci. 2000;917:522-33. doi: 10.1111/j.1749-6632.2000.tb05417.x. PMID 11268380
- [Background] Krishnan N, Thellin O, Buckley DJ, Horseman ND, Buckley AR. Prolactin suppresses glucocorticoid-induced thymocyte apoptosis in vivo. Endocrinology. 2003 May;144(5):2102-10. doi: 10.1210/en.2003-0053. PMID 12697719
- [Background] Leff MA, Buckley DJ, Krumenacker JS, Reed JC, Miyashita T, Buckley AR. Rapid modulation of the apoptosis regulatory genes, bcl-2 and bax by prolactin in rat Nb2 lymphoma cells. Endocrinology. 1996 Dec;137(12):5456-62. doi: 10.1210/endo.137.12.8940371.
- [Background] Buckley AR, Buckley DJ, Leff MA, Hoover DS, Magnuson NS. Rapid induction of pim-1 expression by prolactin and interleukin-2 in rat Nb2 lymphoma cells. Endocrinology. 1995 Dec;136(12):5252-9. doi: 10.1210/endo.136.12.7588268.
- [Background] Hotchkiss RS, Swanson PE, Knudson CM, Chang KC, Cobb JP, Osborne DF, Zollner KM, Buchman TG, Korsmeyer SJ, Karl IE. Overexpression of Bcl-2 in transgenic mice decreases apoptosis and improves survival in sepsis. J Immunol. 1999 Apr 1;162(7):4148-56. PMID 10201940
- [Background] Matera L. Endocrine, paracrine and autocrine actions of prolactin on immune cells. Life Sci. 1996;59(8):599-614. doi: 10.1016/0024-3205(96)00225-1. PMID 8761011
- [Background] Berczi I. Pituitary hormones and immune function. Acta Paediatr Suppl. 1997 Nov;423:70-5. doi: 10.1111/j.1651-2227.1997.tb18376.x. PMID 9401545
- [Background] Buckley AR. Prolactin, a lymphocyte growth and survival factor. Lupus. 2001;10(10):684-90. doi: 10.1191/096120301717164912. PMID 11721694
- [Background] Chikanza IC. Prolactin and neuroimmunomodulation: in vitro and in vivo observations. Ann N Y Acad Sci. 1999 Jun 22;876:119-30. doi: 10.1111/j.1749-6632.1999.tb07629.x. PMID 10415600
- [Background] Fraker PJ, King LE, Laakko T, Vollmer TL. The dynamic link between the integrity of the immune system and zinc status. J Nutr. 2000 May;130(5S Suppl):1399S-406S. doi: 10.1093/jn/130.5.1399S. PMID 10801951
- [Background] Newsholme P, Curi R, Pithon Curi TC, Murphy CJ, Garcia C, Pires de Melo M. Glutamine metabolism by lymphocytes, macrophages, and neutrophils: its importance in health and disease. J Nutr Biochem. 1999 Jun;10(6):316-24. doi: 10.1016/s0955-2863(99)00022-4. PMID 15539305
- [Background] King LE, Osati-Ashtiani F, Fraker PJ. Apoptosis plays a distinct role in the loss of precursor lymphocytes during zinc deficiency in mice. J Nutr. 2002 May;132(5):974-9. doi: 10.1093/jn/132.5.974. PMID 11983824
- [Background] Aleksandrowicz J, Starek A, Moszczynski P. [Effect of selenium on peripheral blood in rats chronically exposed to benzene]. Med Pr. 1977;28(6):453-9. Polish. PMID 609322
- [Background] Szondy Z. The effects of cell number, concentrations of mitogen and glutamine and time of culture on [3H]thymidine incorporation into cervical lymph node lymphocytes stimulated by concanavalin-A. Immunol Lett. 1995 Mar;45(3):167-71. doi: 10.1016/0165-2478(94)00256-q. PMID 7558169
- [Background] Devins SS, Miller A, Herndon BL, O'Toole L, Reisz G. Effects of dopamine on T-lymphocyte proliferative responses and serum prolactin concentrations in critically ill patients. Crit Care Med. 1992 Dec;20(12):1644-9. doi: 10.1097/00003246-199212000-00007. PMID 1458939
- [Background] Van den Berghe G, de Zegher F, Lauwers P. Dopamine suppresses pituitary function in infants and children. Crit Care Med. 1994 Nov;22(11):1747-53. PMID 7956277
- [Background] Van den Berghe G, de Zegher F. Anterior pituitary function during critical illness and dopamine treatment. Crit Care Med. 1996 Sep;24(9):1580-90. doi: 10.1097/00003246-199609000-00024. PMID 8797634
- [Background] Le Saux NM, Sekla L, McLeod J, Parker S, Rush D, Jeffery JR, Brunham RC. Epidemic of nosocomial Legionnaires' disease in renal transplant recipients: a case-control and environmental study. CMAJ. 1989 May 1;140(9):1047-53. PMID 2650836
- [Background] Parra A, Ramirez-Peredo J, Larrea F, Cabrera V, Coutino B, Torres I, Angeles A, Perez-Romano B, Ruiz-Arguelles G, Ruiz-Arguelles A. Decreased dopaminergic tone and increased basal bioactive prolactin in men with human immunodeficiency virus infection. Clin Endocrinol (Oxf). 2001 Jun;54(6):731-8. doi: 10.1046/j.1365-2265.2001.01262.x. PMID 11422107
- [Background] Parra A, Ramirez-Peredo J. The uncoupled couple? Prolactin and CD4 lymphocytes in HIV infection. Med Hypotheses. 1999 Nov;53(5):425-8. doi: 10.1054/mehy.1999.0930. PMID 10616045
- [Background] Ijaiya K, Roth B, Schwenk A. The effects of arginine, insulin and metoclopramide on growth hormone, prolactin and cortisol release in children. Clin Endocrinol (Oxf). 1980 Jun;12(6):589-94. doi: 10.1111/j.1365-2265.1980.tb01380.x. PMID 6994940
- [Background] LL Brunton. Agents affecting gastrointestinal water flux and motility. In Limbird LE Hardman JG, editor, Goodman and Gilman's The Pharmacological Basis of Therapeutics, pages 931-933. McGraw-Hill, New York, 9th edition, 1996.
- [Background] F Shann, editor. Drug Doses. Collective Pty Ltd., Melbourne, 12th edition, 2003.
- [Background] PR Dallman. White blood cells: developmental changes in numbers. In Ruolph CD Rudolph AM, Hoffman JIE, editor, Pediatrics, page 1061. Appleton and Lange, Norwalk CT, 19th edition, 1987.
- [Background] Anonymous. Immunization in special clinical circumstances. In LK Pickering, editor, 2000 Redbook: Report of the Committee of Infectious Diseases, page 59. Academy of Pediatrics, Elk Grove Village, IL, 25th edition, 2000.
- [Background] E.R. Stiehm. Immunologic disorders in infants and children. W.B. Saunders, Philadelphia, PA, 1989.
- [Background] Hotchkiss RS, Tinsley KW, Swanson PE, Schmieg RE Jr, Hui JJ, Chang KC, Osborne DF, Freeman BD, Cobb JP, Buchman TG, Karl IE. Sepsis-induced apoptosis causes progressive profound depletion of B and CD4+ T lymphocytes in humans. J Immunol. 2001 Jun 1;166(11):6952-63. doi: 10.4049/jimmunol.166.11.6952. PMID 11359857
- [Background] Gurevich P, Ben-Hur H, Czernobilsky B, Nyska A, Zuckerman A, Zusman I. Pathology of lymphoid organs in low birth weight infants subjected to antigen-related diseases: a morphological and morphometric study. Pathology. 1995 Apr;27(2):121-6. doi: 10.1080/00313029500169702. PMID 7567136
- [Background] Hotchkiss RS, Chang KC, Swanson PE, Tinsley KW, Hui JJ, Klender P, Xanthoudakis S, Roy S, Black C, Grimm E, Aspiotis R, Han Y, Nicholson DW, Karl IE. Caspase inhibitors improve survival in sepsis: a critical role of the lymphocyte. Nat Immunol. 2000 Dec;1(6):496-501. doi: 10.1038/82741. PMID 11101871
- [Background] Zellweger R, Wichmann MW, Ayala A, Chaudry IH. Metoclopramide: a novel and safe immunomodulating agent for restoring the depressed macrophage immune function after hemorrhage. J Trauma. 1998 Jan;44(1):70-7. doi: 10.1097/00005373-199801000-00006. PMID 9464751
- [Background] Zellweger R, Zhu XH, Wichmann MW, Ayala A, DeMaso CM, Chaudry IH. Prolactin administration following hemorrhagic shock improves macrophage cytokine release capacity and decreases mortality from subsequent sepsis. J Immunol. 1996 Dec 15;157(12):5748-54. PMID 8955229
- [Background] Knoferl MW, Angele MK, Ayala A, Cioffi WG, Bland KI, Chaudry IH. Insight into the mechanism by which metoclopramide improves immune functions after trauma-hemorrhage. Am J Physiol Cell Physiol. 2000 Jul;279(1):C72-80. doi: 10.1152/ajpcell.2000.279.1.C72. PMID 10898718
- [Background] Felmet KA, Hall MW, Clark RS, Jaffe R, Carcillo JA. Prolonged lymphopenia, lymphoid depletion, and hypoprolactinemia in children with nosocomial sepsis and multiple organ failure. J Immunol. 2005 Mar 15;174(6):3765-72. doi: 10.4049/jimmunol.174.6.3765. PMID 15749917
- [Background] Yavagal DR, Karnad DR, Oak JL. Metoclopramide for preventing pneumonia in critically ill patients receiving enteral tube feeding: a randomized controlled trial. Crit Care Med. 2000 May;28(5):1408-11. doi: 10.1097/00003246-200005000-00025. PMID 10834687
- [Background] Brooks WA, Yunus M, Santosham M, Wahed MA, Nahar K, Yeasmin S, Black RE. Zinc for severe pneumonia in very young children: double-blind placebo-controlled trial. Lancet. 2004 May 22;363(9422):1683-8. doi: 10.1016/S0140-6736(04)16252-1. PMID 15158629
- [Background] Fischer Walker C, Black RE. Zinc and the risk for infectious disease. Annu Rev Nutr. 2004;24:255-75. doi: 10.1146/annurev.nutr.23.011702.073054. PMID 15189121
- [Background] Baqui AH, Black RE, El Arifeen S, Yunus M, Zaman K, Begum N, Roess AA, Santosham M. Zinc therapy for diarrhoea increased the use of oral rehydration therapy and reduced the use of antibiotics in Bangladeshi children. J Health Popul Nutr. 2004 Dec;22(4):440-2. PMID 15663177
- [Background] Raqib R, Roy SK, Rahman MJ, Azim T, Ameer SS, Chisti J, Andersson J. Effect of zinc supplementation on immune and inflammatory responses in pediatric patients with shigellosis. Am J Clin Nutr. 2004 Mar;79(3):444-50. doi: 10.1093/ajcn/79.3.444. PMID 14985220
- [Background] Bhatnagar S, Bahl R, Sharma PK, Kumar GT, Saxena SK, Bhan MK. Zinc with oral rehydration therapy reduces stool output and duration of diarrhea in hospitalized children: a randomized controlled trial. J Pediatr Gastroenterol Nutr. 2004 Jan;38(1):34-40. doi: 10.1097/00005176-200401000-00010. PMID 14676592
- [Background] Sazawal S, Black RE, Menon VP, Dinghra P, Caulfield LE, Dhingra U, Bagati A. Zinc supplementation in infants born small for gestational age reduces mortality: a prospective, randomized, controlled trial. Pediatrics. 2001 Dec;108(6):1280-6. doi: 10.1542/peds.108.6.1280. PMID 11731649
- [Background] Darlow BA, Austin NC. Selenium supplementation to prevent short-term morbidity in preterm neonates. Cochrane Database Syst Rev. 2003;2003(4):CD003312. doi: 10.1002/14651858.CD003312. PMID 14583967
- [Background] van den Berg A, van Elburg RM, Westerbeek EA, Twisk JW, Fetter WP. Glutamine-enriched enteral nutrition in very-low-birth-weight infants and effects on feeding tolerance and infectious morbidity: a randomized controlled trial. Am J Clin Nutr. 2005 Jun;81(6):1397-404. doi: 10.1093/ajcn/81.6.1397. PMID 15941893
- [Background] Boelens PG, Houdijk AP, Fonk JC, Puyana JC, Haarman HJ, von Blomberg-van der Flier ME, van Leeuwen PA. Glutamine-enriched enteral nutrition increases in vitro interferon-gamma production but does not influence the in vivo specific antibody response to KLH after severe trauma. A prospective, double blind, randomized clinical study. Clin Nutr. 2004 Jun;23(3):391-400. doi: 10.1016/j.clnu.2003.09.002. PMID 15158303
- [Background] Yalcin SS, Yurdakok K, Tezcan I, Oner L. Effect of glutamine supplementation on diarrhea, interleukin-8 and secretory immunoglobulin A in children with acute diarrhea. J Pediatr Gastroenterol Nutr. 2004 May;38(5):494-501. doi: 10.1097/00005176-200405000-00007. PMID 15097437
- [Background] Leteurtre S, Martinot A, Duhamel A, Gauvin F, Grandbastien B, Nam TV, Proulx F, Lacroix J, Leclerc F. Development of a pediatric multiple organ dysfunction score: use of two strategies. Med Decis Making. 1999 Oct-Dec;19(4):399-410. doi: 10.1177/0272989X9901900408. PMID 10520678
- [Background] Leteurtre S, Martinot A, Duhamel A, Proulx F, Grandbastien B, Cotting J, Gottesman R, Joffe A, Pfenninger J, Hubert P, Lacroix J, Leclerc F. Validation of the paediatric logistic organ dysfunction (PELOD) score: prospective, observational, multicentre study. Lancet. 2003 Jul 19;362(9379):192-7. doi: 10.1016/S0140-6736(03)13908-6. PMID 12885479
- [Background] Doughty LA, Kaplan SS, Carcillo JA. Inflammatory cytokine and nitric oxide responses in pediatric sepsis and organ failure. Crit Care Med. 1996 Jul;24(7):1137-43. doi: 10.1097/00003246-199607000-00012. PMID 8674325
- [Background] Pollack MM, Patel KM, Ruttimann UE. The Pediatric Risk of Mortality III--Acute Physiology Score (PRISM III-APS): a method of assessing physiologic instability for pediatric intensive care unit patients. J Pediatr. 1997 Oct;131(4):575-81. doi: 10.1016/s0022-3476(97)70065-9. PMID 9386662
- [Background] Slota M, Green M, Farley A, Janosky J, Carcillo J. The role of gown and glove isolation and strict handwashing in the reduction of nosocomial infection in children with solid organ transplantation. Crit Care Med. 2001 Feb;29(2):405-12. doi: 10.1097/00003246-200102000-00034. PMID 11246324
- [Background] Leclerc F, Leteurtre S, Duhamel A, Grandbastien B, Proulx F, Martinot A, Gauvin F, Hubert P, Lacroix J. Cumulative influence of organ dysfunctions and septic state on mortality of critically ill children. Am J Respir Crit Care Med. 2005 Feb 15;171(4):348-53. doi: 10.1164/rccm.200405-630OC. Epub 2004 Oct 29. PMID 15516535
- [Background] Klein BS, Perloff WH, Maki DG. Reduction of nosocomial infection during pediatric intensive care by protective isolation. N Engl J Med. 1989 Jun 29;320(26):1714-21. doi: 10.1056/NEJM198906293202603. PMID 2733733
- [Background] Carcillo J, Holubkov R, Dean JM, Berger J, Meert KL, Anand KJ, Zimmerman J, Newth CJ, Harrison R, Willson DF, Nicholson C; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Rationale and design of the pediatric critical illness stress-induced immune suppression (CRISIS) prevention trial. JPEN J Parenter Enteral Nutr. 2009 Jul-Aug;33(4):368-74. doi: 10.1177/0148607108327392. Epub 2009 Apr 14. PMID 19380753
- [Result] Carcillo JA, Dean JM, Holubkov R, Berger J, Meert KL, Anand KJ, Zimmerman J, Newth CJ, Harrison R, Burr J, Willson DF, Nicholson C; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Collaborative Pediatric Critical Care Research Network (CPCCRN). The randomized comparative pediatric critical illness stress-induced immune suppression (CRISIS) prevention trial. Pediatr Crit Care Med. 2012 Mar;13(2):165-73. doi: 10.1097/PCC.0b013e31823896ae. PMID 22079954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: April 2007 - November 2009; Location: Pediatric Intensive Care Unit (PICU)
Pre-assignment Details: Patients were stratified according to immunocompromised status prior to randomization.
Groups:
- Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide: Subjects assigned to this group received zinc (20 mg), selenium (40 mcg ages 1-3 yrs, 100 mcg age 3-5 yrs, 200 mcg age 5-12 yrs, 400 mcg adolescent), and glutamine (0.3 g/kg) each morning, and intravenous metoclopramide (0.2 mg/kg, maximum 10 mg) every 12 hrs.
- Enteral Whey Protein, IV Saline: Subjects assigned to the whey protein group received 0.3 g/kg beneprotein each morning and intravenous saline every 12 hrs.
Period: Overall Study
Arm/Group | Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide | Enteral Whey Protein, IV Saline
Started | 149 | 144
Completed | 149 | 144
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Daily Nutriceutical Supplementation: Subjects assigned to this group received zinc (20 mg), selenium (40 mcg ages 1-3 yrs, 100 mcg age 3-5 yrs, 200 mcg age 5-12 yrs, 400 mcg adolescent), and glutamine (0.3 g/kg) each morning, and intravenous metoclopramide (0.2 mg/kg, maximum 10 mg) every 12 hrs.
- Whey Protein: Subjects assigned to the whey protein group received 0.3 g/kg beneprotein each morning and intravenous saline every 12 hrs.
- Total: Total of all reporting groups
Arm/Group | Daily Nutriceutical Supplementation | Whey Protein | Total
Number analyzed (Participants) | 149 | 144 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 149 | 144 | 293
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.9 (5.6) | 8.4 (5.9) | 8.1 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 79 | 148
  Male | 80 | 65 | 145
Region of Enrollment [Number; unit: participants]
  United States | 149 | 144 | 293
Immune Compromised at Study Entry [Number; unit: Participants] — Patients were classified as immune compromised if they had acquired immunodeficiency syndrome, cancer, transplantation, primary immune deficiency or chronic immune suppressant therapy.
  Participants
    Immune compromised | 14 | 11 | 25
    Immune Competent | 135 | 133 | 268

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study is the Median Time Between Admission to the PICU and Occurrence of Nosocomial Infection or Clinical Sepsis in PICU Patients Who Have Endotracheal Tubes, Central Venous Catheters, or Urinary Catheters.
Time Frame: 48 hours after admission until 5 days after discharged from the PICU
Population: Intention to treat analysis of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Daily Nutriceutical Supplementation | Whey Protein
Number analyzed (Participants) | 149 | 144
Days | 12.1 [9.25 to 32.4] | 13.2 [10.8 to NA] — The upper limit of the 95% confidence interval for median number of days to event in this arm is not calculable due to an insufficient number of participants reaching the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Daily Nutriceutical Supplementation vs Whey Protein; Null hypothesis was equal median time in both arms. Sample size calculated to yield 90% power to detect a significant effect, assuming inverse hazard rate of 1.5 using two-sided logrank test with alpha=0.05. This required recruitment until 263 patients with an event were enrolled (though the study was terminated early for futility by the DSMB); Test type: Superiority or Other; p = 0.29, Log Rank; Two-sided logrank test was used, stratified by immune compromised status at study entry (a factor also used to stratify the study randomization)

2. Secondary Outcome: Rate of Nosocomial Infection or Clinical Sepsis Per 100 Study Days
Time Frame: 48 hours after PICU admission till discharge from PICU
Population: All randomized patients analyzed by intention to treat
Measure: Mean (95% Confidence Interval); unit: Mean number of events per 100 study days
Arm/Group | Daily Nutriceutical Supplementation | Whey Protein
Number analyzed (Participants) | 149 | 144
Mean number of events per 100 study days | 4.99 [4.12 to 5.99] | 4.83 [4.01 to 5.77]
Statistical Analysis 1: Comparison: Daily Nutriceutical Supplementation vs Whey Protein; Null hypothesis of equal event rates in the two study arms; Test type: Superiority or Other; p = 0.81, Rate analysis (see comments); 95% CIs were calculated for rates in each arm, and rates compared between arms, via approach of DR Cox, Biometrika (1953), vol 40, pp. 354-60

3. Secondary Outcome: Antibiotic-free Days
Time Frame: 48 hours after admission until PICU discharge
Population: All randomized patients per intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide | Enteral Whey Protein, IV Saline
Number analyzed (Participants) | 149 | 144
Days | 1 [0 to 5] | 2 [0 to 6]
Statistical Analysis 1: Comparison: Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide vs Enteral Whey Protein, IV Saline; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Incidence of Prolonged Lymphopenia (Absolute Lymphocyte Count Less Than or Equal to 1,000/mm³ for > or Equal to 7 Days)
Description: What is reported is the number of participants with counts qualifying as lymphopenia.
Time Frame: from time of PICU admission till discharge from PICU
Population: All randomized patients (intention to treat analysis)
Measure: Number; unit: participants
Arm/Group | Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide | Enteral Whey Protein, IV Saline
Number analyzed (Participants) | 149 | 144
participants | 5 | 12
Statistical Analysis 1: Comparison: Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide vs Enteral Whey Protein, IV Saline; Test type: Superiority or Other; p = 0.07, Chi-squared

5. Secondary Outcome: All-cause 28-day Mortality Rate.
Time Frame: 28 days after admission to the PICU
Population: This safety outcome was analyzed by treatment received, among a total of 284 children who received treatment and had known 28-day status.
Measure: Number; unit: participants
Arm/Group | Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide | Enteral Whey Protein, IV Saline
Number analyzed (Participants) | 145 | 139
participants | 15 | 8
Statistical Analysis 1: Comparison: Enteral Zinc, Selenium, Glutamine, and IV Metoclopramide vs Enteral Whey Protein, IV Saline; Test type: Superiority or Other; p = 0.16, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 28 days.
Description: For adverse events, denominators reflect Safety Population of those patients receiving each treatment. Therefore, denominators are 148 patients receiving Daily Nutriceutical Supplementation and 139 patients receiving Whey Protein.
Arm/Group | Daily Nutriceutical Supplementation | Whey Protein
Serious Adverse Events (participants affected / at risk) | 73/148 | 70/139
Other Adverse Events (participants affected / at risk) | 119/148 | 112/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Nutriceutical Supplementation (N=148) | Whey Protein (N=139)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 4 (6)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 2 (3)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1)
Cortical blindness (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischemic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Multiple organ failure (General disorders) | 2 (2) | 1 (1)
Withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Nosocomial infection (Infections and infestations) | 43 (73) | 41 (61)
Sepsis (Infections and infestations) | 13 (14) | 20 (29)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase high (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
CSF WBC increased (Investigations) | 0 (0) | 1 (1)
Culture stool positive (Investigations) | 1 (1) | 0 (0)
Culture urine positive (Investigations) | 1 (1) | 0 (0)
Decreased INR (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
PCO2 increased (Investigations) | 0 (0) | 2 (2)
WBC increased (Investigations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute myeloid leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral edema (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral infarct (Nervous system disorders) | 0 (0) | 1 (1)
Choreoathetoid movements (Nervous system disorders) | 0 (0) | 2 (2)
Consciousness decreased (Nervous system disorders) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 1 (1)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Shaking (Nervous system disorders) | 1 (1) | 0 (0)
Acute mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure NOS (Renal and urinary disorders) | 0 (0) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Failure respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Paralysis of diaphragm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Nutriceutical Supplementation (N=148) | Whey Protein (N=139)
Anemia (Blood and lymphatic system disorders) | 9 (10) | 10 (11)
Coagulopathy (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 10 (11) | 10 (10)
Bradycardia (Cardiac disorders) | 17 (19) | 14 (15)
Tachycardia (Cardiac disorders) | 11 (12) | 20 (24)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 7 (8)
Constipation (Gastrointestinal disorders) | 21 (21) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 10 (13)
Emesis (Gastrointestinal disorders) | 19 (25) | 17 (22)
Vomiting (Gastrointestinal disorders) | 6 (7) | 10 (10)
Fever (General disorders) | 13 (13) | 13 (15)
Hyperthermia (General disorders) | 10 (12) | 9 (14)
Hypothermia (General disorders) | 10 (19) | 8 (8)
Pyrexia (General disorders) | 16 (22) | 14 (18)
Nosocomial infection (Infections and infestations) | 8 (9) | 10 (13)
Sepsis (Infections and infestations) | 8 (8) | 7 (11)
BUN increased (Investigations) | 11 (12) | 8 (9)
Blood albumin decreased (Investigations) | 4 (4) | 8 (8)
Blood magnesium decreased (Investigations) | 15 (16) | 10 (11)
Blood phosphorus decreased (Investigations) | 13 (17) | 13 (14)
Blood potassium decreased (Investigations) | 11 (11) | 11 (13)
Blood sodium decreased (Investigations) | 6 (6) | 7 (8)
Hematocrit decreased (Investigations) | 12 (13) | 10 (10)
Hemoglobin decreased (Investigations) | 13 (14) | 10 (17)
Lipase increased (Investigations) | 13 (14) | 5 (5)
Oxygen saturation decreased (Investigations) | 18 (20) | 13 (15)
PCO2 increased (Investigations) | 3 (5) | 8 (11)
Platelets decreased (Investigations) | 6 (7) | 7 (8)
Acidosis (Metabolism and nutrition disorders) | 5 (7) | 8 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (27) | 19 (21)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 8 (10)
Hypernatremia (Metabolism and nutrition disorders) | 11 (12) | 8 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 8 (10)
Hypokalemia (Metabolism and nutrition disorders) | 26 (30) | 27 (41)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (6) | 7 (12)
Hyponatremia (Metabolism and nutrition disorders) | 7 (8) | 11 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 8 (9)
Seizure (Nervous system disorders) | 3 (4) | 7 (7)
Agitation (Psychiatric disorders) | 18 (18) | 18 (19)
Oliguria (Renal and urinary disorders) | 8 (9) | 8 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 17 (20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 9 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (16)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 13 (21)
Stridor (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (14)
Skin breakdown (Skin and subcutaneous tissue disorders) | 7 (11) | 8 (15)
Hypertension (Vascular disorders) | 23 (24) | 16 (19)
Hypotension (Vascular disorders) | 32 (37) | 32 (39)

LIMITATIONS AND CAVEATS:
The Data Safety Monitoring Board met on November 30, 2009. Interim analysis of the first 273 patients was presented. Per the Board's recommendations, the study was terminated based on futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No